CLINICAL TRIAL: NCT03894098
Title: High Ankle Block Versus Regional Block for Acute Pain Control After Ankle Surgery: A Prospective Randomized Controlled Study
Brief Title: High Ankle Block Versus Regional Block for Acute Pain Control After Ankle Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Low interest.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Glenn G. Shi, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-002398
Record Dates: First submitted 2019-03-27; First posted 2019-03-28 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Ankle Surgery
Keywords: nerve block
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single shot regional popliteal and saphenous block (Active Comparator): Standard of care traditional single shot popliteal / saphenous regional block for acute pain control after elective ankle surgery
  Interventions: Procedure: Nerve block
- High ankle block (Experimental): High ankle block for acute pain control after elective ankle surgery
  Interventions: Procedure: Nerve block

INTERVENTIONS:
Procedure: Nerve block — High ankle nerve block

SUMMARY:
Researchers are trying to determine if a high ankle block during ankle surgery provides the same pain relief as the standard regional block.

DETAILED DESCRIPTION:
Participants scheduled for elective ankle surgery will be randomized to have either a high ankle nerve block or a regional nerve block. Pain levels after surgery will be assessed to determine whether one type of block provides better pain relief compared to the other.

ELIGIBILITY:
Inclusion Criteria

* Adults undergoing elective foot and ankle surgery
* Adults ≥18 years, intact presurgical peripheral sensation based on 5.07 monofilament testing, foot and ankle surgery

Exclusion Criteria

* Presurgical neurologic discrepancies (peripheral neuropathy, radiculopathy)
* Complex regional pain syndrome
* peripheral nerve surgery
* Surgery above the level of the tibiotalar joint
* Narcotic dependency
* Anyone unable to receive a high ankle block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Change in pain score | 24 hours, 48 hours, 72 hours
  Measured using Defense and Veterans Pain Scale (lowest score of 0 = No pain and 10 = As bad as it could be, nothing else matters)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn G Shi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials